CLINICAL TRIAL: NCT00952068
Title: A Pharmacodynamic/Pharmacokinetic Study to Determine the Onset of Analgesic Effect and Plasma Levels of Tramadol in Patients With Acute Low Back Pain Receiving a Single 200 mg Dose of Tramadol Contramid® Once-a-Day
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT2-002; NCT00952068 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2009-04-16; First posted 2009-08-04 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Acute Low Back Pain
Keywords: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tramadol Contramid® OAD 200mg (Experimental): 1 Tramadol Contramid® OAD 200mg tablet daily.
  Interventions: Drug: Tramadol Contramid® OAD 200mg

INTERVENTIONS:
Drug: Tramadol Contramid® OAD 200mg — 1 Tramadol Contramid® OAD 200mg tablet daily.

SUMMARY:
The primary objective of this study is to determine the time of onset of analgesic effect of Tramadol Contramid® Once-A-Day (OAD) in acute low back pain. Secondary objectives include determining the relationship between analgesic effect and plasma levels for Tramadol Contramid® OAD and to examine safety after single dose administration of 200 mg of Tramadol Contramid® OAD.

ELIGIBILITY:
Inclusion Criteria:

* Males or females in generally good health aged 18-80 years with acute low back pain are eligible for this study.
* Patients must have pain of moderate to severe intensity on the patient rating of pain intensity scale without analgesia.
* Oral and written language comprehension at a level sufficient to comply with the protocol and complete study-related materials.
* Must have signed and dated an REB-approved written Informed Consent form which was also signed and dated by the Investigator prior to study participation.

Exclusion Criteria:

* Known history or symptoms suspicious of:

  * Spinal fracture
  * Cancer (i.e. constitutional symptoms such as recent unexplained chills or weight loss)
  * Spinal infection (e.g. IV drug abuse, immunosuppression)
* Cauda equina syndrome
* Spina bifida
* Foot drop
* Spinal surgery within 1 year of study entry
* Body Mass Index (BMI) > 37
* Continuous chronic back pain
* More severe pain in a region other than the lower back
* Treatment of the back pain with non-pharmacological therapy (e.g. acupuncture chiropractic adjustment, Transcutaneous Electrical Nerve Stimulation, physiotherapy etc.) in the 3 weeks prior to study entry
* Use of any sedative hypnotics, topical preparations/medications and anaesthetics or muscle relaxants within 5 half-lives of the dose of study medication
* Use of any analgesic within 6 hours of the dose of study medication. In rare cases, if a patient is in moderate to severe pain despite having taken a short-acting analgesic and if at least 2 hours have passed since the dose of short-acting analgesic, the patient may be entered.
* A major illness, requiring hospitalisation during the 3 months before commencement of the screening period
* Unwillingness to stop taking pain medication other than the study medication
* Previous failure of treatment with tramadol or discontinuation of treatment with tramadol due to adverse events
* Treatment within the last 3 weeks with any of the following medications: monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds (e.g. cyclobenzaprine, promethazine); neuroleptics; selective serotonin reuptake inhibitors (SSRIs); serotonin-norepinephrine reuptake inhibitors (SNRIs) or any other drug that reduces seizure threshold
* Treatment with another investigational agent within the last 30 days
* History of seizure disorder other than Infantile Febrile Seizures
* Previous or current opioid dependency
* Bowel disease causing malabsorption
* Pregnant or lactating women
* Known significant liver disease or symptoms of significant liver disease
* Known significant renal disease or symptoms of significant renal disease
* Current or past substance abuse or dependence, other than nicotine
* Allergy to tramadol or any structurally similar drugs (e.g. opiates)
* Any other condition that, in the opinion of the Investigators, would adversely affect the patient's ability to complete the study or its measures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

REFERENCES:
- [Result] Sarbu A, Radulescu F, Robertson S, Bouchard S. Onset of analgesic effect and plasma levels of controlled-release tramadol (Tramadol Contramid once-a-day) 200-mg tablets in patients with acute low back pain. J Opioid Manag. 2008 Sep-Oct;4(5):285-92. doi: 10.5055/jom.2008.0032. PMID 19070266
- See also: Approved labelling — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Label_ApprovalHistory

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Contramid® Once-A-Day (OAD): Single dose 200 mg of Tramadol Contramid® Once-A-Day (OAD)
Period: Overall Study
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Started | 47
Completed | 40
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 10
Region of Enrollment [Number; unit: participants]
  Romania | 47

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Perceptible Pain Relief
Description: Kaplan-Meier estimates of time to perceptible pain relief. Patients who discontinued or completed the study without perceptible pain relief were censored at the time point of their last pain intensity score. A confidence interval for the median survival time was calculated.
Time Frame: 6 hours
Population: Full analysis population: includes all patients who received the dose of study medication and who had at least one pharmacodynamic assessment during the dosing phase.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Number analyzed (Participants) | 46
minutes | 47 [40 to 51]

2. Secondary Outcome: Patient Rating of Pain Intensity at Onset of Perceptible Pain Relief, 3 Hours and 6 Hours Post Dose
Description: Pain intensity rating at baseline, time of onset of perceptible pain relief, 3 hours and 6 hours post-dose or if the patient discontinued earlier. "What is your current level of pain intensity?" 0=none, 1=mild, 2=moderate, 3=severe. Missing data were imputed using Last Observation Carried Forward (LOCF).
Time Frame: Baseline, 3 hours post-dose, 6 hours post-dose, time of onset of perceptible pain relief
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Number analyzed (Participants) | 46
participants
  Baseline, moderate pain | 34
  Baseline, severe pain | 12
  Onset of perceptible pain relief, no pain | 4
  Onset of perceptible pain relief, mild pain | 23
  Onset of perceptible pain relief, moderate pain | 19
  3 hours post-dose, no pain | 12
  3 hours post-dose, mild pain | 25
  3 hours post-dose, moderate pain | 9
  6 hours post-dose, no pain | 24
  6 hours post-dose, mild pain | 20
  6 hours post-dose, moderate pain | 2

3. Secondary Outcome: Patient Rating of Pain Relief at Onset of Perceptible Pain Relief, 3 Hours and 6 Hours Post Dose
Description: Pain relief rating at time of onset of perceptible pain relief, 3 hours and 6 hours post-dose or if the patient discontinued earlier. " How would you rate the pain relief the study medication has given you?" ranging from 0=none to 4=complete relief. Missing data were imputed using Last Observation Carried Forward (LOCF).
Time Frame: 3 hours post-dose, 6 hours post-dose, at time of onset of perceptible pain relief
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Number analyzed (Participants) | 46
participants
  Onset of perceptible pain relief, no pain relief | 1
  Onset of perceptible pain relief, a little relief | 16
  Onset of perceptible pain relief, moderate relief | 9
  Onset of perceptible pain relief, a lot of relief | 16
  Onset of perceptible pain relief, complete relief | 4
  3 hours post-dose, no pain relief | 2
  3 hours post-dose, a little relief | 3
  3 hours post-dose, moderate relief | 12
  3 hours post-dose, a lot of relief | 17
  3 hours post-dose, complete relief | 12
  6 hours post-dose, no pain relief | 1
  6 hours post-dose, a little relief | 2
  6 hours post-dose, moderate relief | 1
  6 hours post-dose, a lot of relief | 18
  6 hours post-dose, complete relief | 24

4. Secondary Outcome: Plasma Levels of Tramadol at 0 Hour (Baseline), Onset of Perceptible Pain Relief, 3 Hours and 6 Hours Post-dose
Description: PK samples were drawn at the end of the Screening Phase, at the onset of perceptible pain relief, at 3 hours and at 6 hours post-dose or if the patient discontinues early. PK samples were always drawn after the completion of the patient ratings of pain relief and of pain intensity scales. They were processed in a central laboratory and the plasma levels of tramadol were collected.
Time Frame: Baseline, time of onset of perceptible pain relief, 3 hours post-dose, 6 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Number analyzed (Participants) | 46
ng/ml
  0 hour | 5.17 (1.55)
  Onset of perceptible pain relief | 56.10 (37.61)
  3 hours post-dose | 176.34 (48.68)
  6 hours post-dose | 187.98 (67.03)

5. Secondary Outcome: Number of Participants With Adverse Events
Description: All adverse events reported during treatment with study drug were considered and reported as treatment emergent adverse events (TEAE) whether or not medication for this adverse event was required by the participant and were summarized in the same table.
Time Frame: 6 hours
Population: Safety population: includes all patients who received the dose of the study medication.
Measure: Number; unit: participants
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Number analyzed (Participants) | 47
participants
  Patients with at least one TEAE | 23
  Patients with at least one severe TEAE | 5
  Patients with at least one SAE | 0
  Patients with at least 1 possibly drug related AE | 23
  Patients with at least one TEAE requiring therapy | 3

ADVERSE EVENTS:
Arm/Group | Tramadol Contramid® Once-A-Day (OAD)
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 23/47
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol Contramid® Once-A-Day (OAD) (N=47)
Somnolence (Nervous system disorders) | 14 (15)
Dizziness (Nervous system disorders) | 8 (12)
Nausea (Gastrointestinal disorders) | 8 (12)
Vomiting NOS (Not Otherwise Specified) (Gastrointestinal disorders) | 5 (10)
Headache NOS (Not Otherwise Specified) (Nervous system disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Bradychardia NOS (Not Otherwise Specified) (Cardiac disorders) | 2 (2)
Sweating increased (Skin and subcutaneous tissue disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 30 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified or delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information.